CLINICAL TRIAL: NCT01914575
Title: Dipole Density Right (and Left) Atrial Mapping and Assessment of Therapy In Complex Supraventricular Tachycardia
Brief Title: Dipole Density Mapping of Right and Left Atrial Supraventricular Tachycardia
Acronym: DDRAMATIC-SVT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Site never got up and running due to institutional issues
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-SVT-003
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Dipole Density Mapping (Experimental)
  Interventions: Device: Mapping with the Acutus Medical System followed by Ablation

INTERVENTIONS:
Device: Mapping with the Acutus Medical System followed by Ablation

SUMMARY:
Use of dipole density mapping to identify activation in complex supraventricular tachycardias

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 75 years
2. scheduled for ablation of atypical atrial flutter or paroxysmal atrial fibrillation
3. able and willing to give informed consent

Exclusion Criteria:

1. implanted prosthetic, artificial, or repaired cardiac valves in the chamber being mapped, permanent pacemaker or ICD leads in the chamber being mapped, and/or hypercoagulopathy or an inability to tolerate anticoagulation .
2. myocardial infarction within the prior two months
3. cardiac surgery within the prior three months
4. intracardiac thrombus
5. clinically significant tricuspid valve regurgitation or stenosis
6. any cerebral ischemic event in the prior six months
7. pregnant or nursing
8. currently enrolled in any other clinical investigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01-22 (Estimated); Primary Completion 2016-05-16 (Actual); Study Completion 2016-05-16 (Actual)

PRIMARY OUTCOMES:
The number of patients with device-related complications | 7 days
The number of patients for which activation maps can be created | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: David Keane, MD, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (1):
- St. Vincent's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No